CLINICAL TRIAL: NCT05034510
Title: A Double-Blind Randomized Crossover Comparison Of Short Pulse Width Versus Low Frequency For Axial Symptoms In Subthalamic Nucleus Deep Brain Stimulation (DBS)-Implanted Parkinson's Disease
Brief Title: Short Pulse Width Versus Low Frequency DBS in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 203/2019/Disp/AOUFe
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-05

CONDITIONS: Parkinson's Disease
Keywords: DBS; Parkinson's disease; low frequency; short pulse width; axial symptoms
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Low frequency 80 Hz then short pulse width 30 usec stimulation (Active Comparator): Each participant will undergo to low frequency stimulation for 4 weeks, then will switch to short pulse width stimulation paradigm for 4 weeks according to the crossover design.
  Interventions: Device: Deep Brain Stimulation
- Short pulse width 30 usec then low frequency 80 Hz stimulation (Active Comparator): Each participant will undergo to short pulse width stimulation paradigm for 4 weeks, then will switch to low frequency for 4 weeks according to the crossover design.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — modification in stimulation parameters

SUMMARY:
The aim is to compare the effect of reducing the conventional pulse width or frequency of stimulation for axial symptoms occurring after Subthalamic nucleus Deep Brain Stimulation (STN DBS) treatment. The participants will be assessed with chronic stimulation with conventional stimulation parameters, namely 60 us and 130 Hz, and after random allocation to short pulse width (30 us) or low frequency (80 Hz).

DETAILED DESCRIPTION:
STN-DBS implanted patient frequently develop axial symptoms, such as gait and speech disorders, after this surgical procedure, which dampens long-term quality of life of Parkinson's disease patients. The pathogenesis is not completely understood, as it could be either due to a long-term stimulation side effect or a symptom with later onset in disease progression which is not well controlled with actual stimulation program. In case of freezing of gait onset in STN-DBS, literature suggest reducing stimulation frequency. Although, low pulse width is a promising option to tackle speech disorders after STN implant, it is not known its potential therapeutic potential on freezing of gait.

The aim of this investigation is to compare the effect of low frequency and short pulse width stimulation in patients, who develop axial symptoms during long-term follow-up in chronic conventional STN DBS.

As per protocol, participants will be assessed at baseline with chronic standard stimulation parameters (60 us and 130 Hz) then they will be randomly allocated either to a low-frequency (80Hz) or a low-pulse arm (30 us). The study is designed such that after scheduled re-assessment the participant will be switched from low frequency arm to short pulse width and vice versa according to the crossover nature of protocol design. Both the rating investigator and the participant are blinded to the allocation, whereas an unblinded investigator will modify the parameters according to allocation arm.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Subthalamic Nucleus Deep Brain Stimulation with chronic conventional stimulation at 60 usec and 130 Hz for at least 3 months
* Movement Disorder Society UPDRS part III 3.11 >1
* Freezing of Gait Questionnaire item-3 >1
* Movement Disorder Society UPDRS part III 3.1 >1
* Montreal Cognitive Assessment > 26
* No psychiatric disorders
* All patients will be ≥ 18 years of age
* Documented informed consent

Exclusion Criteria:

* no documented informed consent
* axial disorders not related to Parkinson's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Freezing of gait incidence reduction | 4 weeks
  change of freezing of gait incidence as measured by Freezing of Gait Questionnaire item-3
Improvement of freezing ratio | 4 weeks
  change in freezing ratio

SECONDARY OUTCOMES:
reduction of freezing of gait duration | 4 weeks
  change of composite measure from item-4, item-5 and item-6 of Freezing of Gait Questionnaire
improvement in speech quality | 4 weeks
  change in Movement Disorder Society UPDRS item 3.1

CONTACTS AND LOCATIONS:
Overall Officials: Mariachiara Sensi, PhD, Principal Investigator — Azienda Ospedaliero Universitaria di Ferrara
Locations (1):
- University Hospital of Ferrara - Arcispedale Sant'Anna, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No